CLINICAL TRIAL: NCT02181946
Title: An Open-label Study in HIV+ Patients to Determine the Effects of Nevirapine (VIRAMUNE®) on the Steady State Pharmacokinetics of Fluconazole (DIFLUCAN®)
Brief Title: Effects of Nevirapine on the Steady State Pharmacokinetics of Fluconazole in HIV Positive Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1361
Record Dates: First submitted 2014-07-02; First posted 2014-07-08 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Fluconazole; Nevirapine

ARMS (1):
- Fluconazole with and without Nevirapine (Experimental)
  Interventions: Drug: Fluconazole; Drug: Nevirapine

INTERVENTIONS:
Drug: Fluconazole
Drug: Nevirapine

SUMMARY:
The purpose of this study was to determine the effects of nevirapine on the steady state pharmacokinetics of fluconazole and to assess the steady-state pharmacokinetics of nevirapine when given in combination with fluconazole.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients between the ages of 18 and 65 years who are seropositive for HIV-1 antibody by an ELISA test and confirmed by an alternative method, e.g. Western Blot
* CD4 + cell count ≥ 100 cells/mm3
* Patients who meet the following laboratory parameters

  * Granulocyte count > 1000 cells/mm3
  * Hemoglobin > 9.0 g/dl (men and women)
  * Platelet count > 75,000 cells/mm3
  * Alkaline phosphatase < 3.0 times the upper limit of normal
  * Aspartame Transaminase (AST) and Alanine Transaminase (ALT) < 3.0 times the upper limit of normal
  * Total bilirubin < 1.5 times the upper limit of normal
* Female patients of childbearing potential must be willing to use a reliable form of contraception which must include a medically approved from of barrier contraception
* Patients able to provide written informed consent and comply with study requirements

Exclusion Criteria:

* Female patients who are pregnant or breast-feeding
* Seated systolic blood pressure below 100 mmHg, or greater than 160 mmHg, and/or heart rate less than 50 or greater than 100 beats/min
* History of drug allergy or known drug hypersensitivity
* Patients receiving any investigational drug, antineoplastic agent or radiotherapy other than local skin radiotherapy treatment within 12 weeks before starting study medication
* Patients requiring systemic treatment with corticosteroids or drugs known to be hepatic enzyme inducers or inhibitors within 28 days of study entry (Study Day 1). Such substances in these categories include: macrolide antibiotics (e.g. erythromycin, clarithromycin, azithromycin, dirithromycin), azole antifungals (e.g. itraconazole), rifabutin and phenytoin
* Patients requiring systemic treatment with CYP3A4 (cytochrome P450 3A4) substrates such as terfenadine, astemizole, cisapride, triazolam and midazolam during the course of the trial
* Use of protease inhibitors or non-nucleoside reverse transcriptase inhibitors within 28 days of Study Day 1 or during the trial
* Patients with a current history of intravenous drug abuse, alcohol or substance abuse (within the last year)
* History of any clinically important disease including hepatic, renal, cardiovascular or gastrointestinal disease
* Patients with malabsorption, severe chronic diarrhea or patients unable to maintain adequate oral intake

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-05; Primary Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Maximum concentration of the analyte in plasma (Cmax) | up to day 40
Minimum concentration of the analyte in plasma (Cmin) | up to day 40
Area under the plasma concentration time curve over the dosing interval (AUCτ) | up to day 40

SECONDARY OUTCOMES:
Time of Cmax (Tmax) | up to day 40
Oral clearance (Cl/F) | up to day 40
Number of patients with adverse events | up to 40 days
Number of patients with abnormal changes in laboratory parameters | up to day 40
Number of patients with clinically significant changes in vital signs | up to day 39